CLINICAL TRIAL: NCT00308945
Title: Influence of Travoprost 0.004% and Latanoprost 0.005% on Retinal Vascular Diameter and Choroidal Blood Flow in Glaucoma Patients
Brief Title: Influence of Prostaglandins on Ocular Blood Flow in Glaucoma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Selim Orgul, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 003-ZAC-2004-001
Record Dates: First submitted 2006-03-29; First posted 2006-03-30 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Open-Angle Glaucoma
Keywords: Glaucoma; Blood flow; Choroid; Retina; Prostaglandin analogues
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Travoprost; Pharmaceutical Preparations; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): cross-over comparison of two substances
  Interventions: Drug: latanoprost 0.005% (drug)
- 1 (Experimental)
  Interventions: Drug: travoprost 0.004% (drug)

INTERVENTIONS:
Drug: travoprost 0.004% (drug) — local drop application
  Arms: 1
Drug: latanoprost 0.005% (drug) — local drop application
  Arms: 2

SUMMARY:
Vasoactivity of topical drugs may be of prognostic relevance in glaucoma. There is very little information for a major class, the prostaglandin analogues with regard to this aspect. The purpose of this study is to compare the effect of travoprost 0.004% and latanoprost 0.005% on choroidal blood flow and retinal vascular diameter in glaucoma patients. After washout of current topical medication, intraocular pressure (IOP) in both eyes (Goldmann applanation tonometry), choroidal blood flow (laser Doppler flowmetry) and retinal vessel diameter (Retinal Vessel Analyzer) in one randomly selected eye will be measured at baseline, after two weeks and after 4 weeks of treatment with travoprost or latanoprost QD, in a randomized, double masked 2-way cross-over study in 20 open angle glaucoma patients.

DETAILED DESCRIPTION:
Background Glaucoma is a leading cause of blindness worldwide. Chronic primary open-angle glaucoma is the most common form among Caucasian patients. The key feature of glaucoma is damage to the optic nerve head, which is not necessarily related to an increase in intraocular pressure (IOP). The actual therapeutic armamentarium for glaucoma includes miotics, beta-blockers, alpha-adrenergic agonists, oral and topical carbonic anhydrase inhibitors, and prostaglandin analogues, the latter being the latest addition to the armamentarium and the most potent topical IOP lowering drugs. Besides IOP, ocular blood flow alterations have been incriminated in glaucoma. Hence, it is of relevance to assess the effect of anti-glaucomatous drugs on ocular blood flow.

Rationale of the study Vasoactivity of topical drugs may be of prognostic relevance in glaucoma. There is very little information for a major class, the prostaglandin analogues with regard to this aspect. The vascular activity of two prostaglandin analogues, travoprost 0.004% and latanoprost 0.005%, which are already on the Swiss market, will be tested.

Study objectives Primary Objective: To assess the effect of two prostaglandin analogues, travoprost 0.004% and latanoprost 0.005% on choroidal blood flow in primary open-angle glaucoma patients.

Secondary Objective: To assess the effect of travoprost 0.004% and latanoprost 0.005% on retinal vascular diameter in primary open-angle glaucoma patients.

Investigational plan Primary open-angle-glaucoma patients will be assessed regarding inclusion/exclusion criteria. After a washout of current topical medication (beta-blockers and prostaglandin analogues: 4 weeks; topical carbonic anhydrase inhibitors and alpha-agonists: 2 weeks; Pilocarpine: 1 week), half of the patients (17 patients) will be treated with travoprost 0.004% for 1 month while the other 17 patients will be treated with latanoprost 0.005% for the same duration. Efficacy and safety variables will be assessed at baseline, after 2 weeks, and after 1 month of treatment. After this first period, the patients will be washed out for 4 weeks and baseline efficacy and safety parameters will be obtained. Afterwards, the patients will be treated with the other compound. Again, efficacy and safety variables will be assessed after 2 weeks and after 1 month of treatment.

Design Single center, randomized, double masked 2-way cross-over design. Randomization The patients will be divided in two groups, and each group will alternatively be started with either travoprost 0.004% or latanoprost 0.005%. Recruitment and management will be carried out by a study nurse masked to baseline blood flow measurement results. Masking and randomization procedures will be entrusted to Alcon PHARMACEUTICAL AG. The drug products for this study will be prepared by the following procedure: Each product will be labeled during independent labeling operations. For this study four different products will have to be labeled: travatan medicin A, travatan medicin B, xalatan medicin A and xalatan medicin B. Each labeling operation will start and end with a line clearance procedure and each labeling order will be 100% inspected by a person that is independent from the person who will do the labeling. On each label the patient number will indicated. The labeling order will be initiated by using the randomization list that indicates which product has to be labeled for which patient. The randomization sequence will be pulled from a uniform distribution with an arbitrary seed (Randomization Performed with SAS 8.2 on NT using RANUNI [seed]). During each independent labeling operation also the disclosure labels will be provided with the same patient number than indicated on the open label. After release of each independent labeling procedure, the assembly of the packaging of two carton boxes in an assembly carton box will start for each patient. The assembly box will also be also labeled with patient number/investigator number and protocol number. Release of the labeled samples will always be done by an independent QA department.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling two out of three of the following criteria in one or both eyes: a) typical glaucomatous disc, b) visual field damage (a cluster of three points (except rim points) in at least one hemifield reduced by 5 dB or greater and including at least one point reduced by 10 dB or greater; a cluster of two points reduced by 10 dB or greater; or three adjacent points on the nasal horizontal meridian that differed by 5 dB or greater from their mirror points on the opposite side of the meridian), c) intraocular pressure above 21 mm Hg at least at one occasion after washout. No closed iridocorneal angles, evidence of secondary glaucoma, pseudoexfoliation, pigmentary dispersion, or any form of retinal or neuroophthalmologic disease that could result in visual field defects. No history of drug or alcohol abuse.

Exclusion Criteria:

* Best corrected visual acuity worse than 2/10 in either eye < 0.2 Snellen. Inadequate transparency of ocular media as defined by physical examination. Severe central field loss defined as a sensitivity < 10dB in at least 2 of the 4 visual field test points closest to the point of fixation. Any abnormality which in the physician's view would prevent reliable applanation tonometry or LDF of both eyes, including an ametropia >3 dpt. History of chronic or recurrent severe inflammatory eye disease such as scleritis or uveitis. History of ocular trauma or intraocular surgery within the past 6 months. History of infection or inflammation within the past 3 months. History of clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy or retinal detachment. A known hypersensitivity to the compounds tested. Need for any concomitant medications that may interfere with the evaluation of ocular blood flow. Variability > 30 % during Laser Doppler Flowmetry (sample of 6 measurements) in both eyes. Pregnancy, breastfeeding, or women in childbearing age without adequate contraception.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-11; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
effect on choroidal blood flow | baseline - 2 weeks - 4 weeks

SECONDARY OUTCOMES:
effect on retinal vascular diameter | baseline - 2 weeks - 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgul, MD, Principal Investigator — University Eye Clinic Basel
Locations (1):
- University Eye Clinic, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- See also: Related Info — http://www.unispital-basel.ch/augenklinik.php